CLINICAL TRIAL: NCT06571019
Title: A Randomized Controlled Trial (RCT) Evaluating the Effects of Cool Roofs on Health Outcomes Using Smartwatches in Niue
Brief Title: Assessing the Effect of Cool Roofs on Health Using Smartwatches in Niue
Acronym: REFLECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aditi Bunker (Other)
Collaborators: Heidelberg University (Other); London School of Hygiene and Tropical Medicine (Other); Rutgers University (Other); Secretaría de Educación Pública, México (Other Government); University of Ouagadougou, Burkina Faso (Other); Indian Institute of Public Health, India (Other); Labfront (Industry); Cognifit (Unknown); Resene (Industry); Habitat for Humanity (Other); The Tindall Foundation (Other); Pacific Community (Other); Wellcome Trust (Other)
Responsible Party: Sponsor-Investigator, Aditi Bunker, Co-Principal Investigator, University of Auckland, New Zealand
Organization: University of Auckland, New Zealand (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3728161; 226745/Z/22/Z (Other Grant/Funding Number: Wellcome Trust UK)
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Heart Rate; All-day Steps; Distance Walked; Active Minutes; Moderate-intensity Activity Minutes; Vigorous-intensity Activity Duration; Sleep Quantity; Time in Sleep Stages; Awake Duration; Sleep Score
Keywords: Hot Temperature; Humidity; Housing; Wearable; Smartwatch; Heart rate; Cardiovascular; Physical activity; Sleep; Cool roof; Heat stress
MeSH Terms: conditions — Motor Activity; Heat Stress Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Trial participants will be aware of the intervention to which they have been allocated, and the research fieldworkers will be aware of the intervention allocation. The trial steering committee members and trial statistician will remain blinded until the end of trial period and data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Households will receive sunlight reflecting 'cool roof' coating on their roofs.
  Interventions: Other: Cool roof
- Control (No Intervention): No cool roof application. Households will keep their original roofing for the duration of the trial.

INTERVENTIONS:
Other: Cool roof — Cool roofs are a heat-reflecting material that can be applied to existing household roofing in the form of a liquid-applied membrane. Cool roofs work by increasing solar reflectance (the ability to reflect the visible wavelengths of sunlight, reducing heat transfer to the surface) and thermal emittance (the ability to radiate absorbed solar energy) thereby reducing the amount of heat transferred into the home.
  Arms: Intervention

SUMMARY:
Ambient air temperatures in the Pacific have broken record highs in 2024. Solutions are needed to build heat resilience in communities and adapt to increasing heat from climate change. Sunlight-reflecting cool roof coatings may passively reduce indoor temperatures and energy use to protect home occupants from extreme heat. Occupants living in poor housing conditions in the Pacific are susceptible to increased heat exposure.

Heat exposure can instigate and worsen numerous physical, mental and social health conditions. The worst adverse health effects are experienced in communities that are least able to adapt to heat exposure. By reducing indoor temperatures, cool roof use may promote heart health, sleep and physical activity in household occupants.

The long-term research goal of the investigators is to identify viable passive housing adaptation technologies with proven health benefits to reduce the burden of heat stress in communities affected by heat in Niue. To meet this goal, the investigators will conduct a randomized controlled trial to establish the effects of cool roof use on heart rate, sleep and physical activity in Niue.

DETAILED DESCRIPTION:
Increasing heat exposure from climate change is causing and exacerbating heat-related illnesses in millions worldwide - particularly in low-resource settings. June 2024 was the 13th consecutive hottest month on record globally - shattering previous records. Heat exposure can instigate and worsen health conditions, including cardiovascular, metabolic, endocrine and respiratory disease, heat-related illnesses, pregnancy complications, and mental health conditions. Adaptation is essential for protecting people from increasing heat exposure. The built environment, especially homes, is ideal for deploying interventions to reduce heat exposure and accelerate adaptation efforts. However, there currently is a lack of evidence on a global scale - generated through empirical studies - guiding the uptake of interventions to reduce heat stress in low-resource settings.

Pacific Islands and other small island developing states are among the most vulnerable to the adverse impacts of climate change and are likely to experience increases in ambient air temperature over the coming decades. People in Niue are exposed to heat and humidity year-round. The Pacific Islands have a large burden of non-communicable diseases (NCDs), with nearly three-quarters of deaths due to NCDs. The combined burden of heat and NCDs places Pacific Island populations at greater risk of adverse health effects from heat extremes.

Sunlight-reflecting cool roof coatings passively reduce indoor temperatures and lower energy use, offering protection to home occupants from extreme heat. The investigators therefore aim to conduct a randomized controlled trial investigating the effects of cool roofs on heart rate, sleep and physical activity using smartwatches in Niue.

The trial will quantify whether cool roofs are an effective passive home cooling intervention with beneficial health effects for vulnerable populations in Niue. Findings will inform regional and global policy responses on scaling cool roof implementation to protect people from increasing heat exposure driven by climate change.

ELIGIBILITY:
Inclusion Criteria:

Participant criteria:

* Consenting adult aged 18 years and over.
* Expected to be available to participate in the study for at least nine months in the next 12 months.
* Willing and able to wear a smartwatch.

Household criteria:

* House has a metal roof.
* House is single-story.

Exclusion Criteria:

Participant criteria:

* One participant per household
* Does not have a smartphone with an internet connection that can connect to the smartwatch.

Household criteria:

* Unstable house structure that does not permit the application of cool roof materials.
* Inaccessible by the research team.
* Significant roof damage defined as any penetrative roof defect that results in a hole in the roof OR over 25% of the roof rusted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  Heart rate in beats per minute measured at 15-second intervals using Garmin Vivosmart 5 devices.

SECONDARY OUTCOMES:
All-day steps | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The number of steps measured daily using Garmin Vivosmart 5 devices.
Active minutes | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The total number of minutes of active exercise daily using Garmin Vivosmart 5 devices.
Distance walked | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The total distance walked daily using Garmin Vivosmart 5 devices.
Moderate-intensity activity minutes | MeasuSmartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at barements will be taken continuously for 12 months. Participants will be asked to wear their smartwatch for at least two weeks every month.
  The total number of minutes of moderate-intensity activity daily using Garmin Vivosmart 5 devices.
Vigorous-intensity activity duration | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The total number of minutes of vigorous-intensity activity daily using Garmin Vivosmart 5 devices.
Sleep quantity | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The number of hours spent asleep each night using Garmin Vivosmart 5 devices.
Time in sleep stages | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The number of hours spent in sleep stages each night using Garmin Vivosmart 5 devices.
Awake duration | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The number of hours spent awake during sleep time each night using Garmin Vivosmart 5 devices.
Sleep score | Smartwatches will be worn for two consecutive weeks per month. Eight measurement points will be taken: one at baseline and seven over 12 months, covering three consecutive hottest months and four alternate months.
  The Garmin sleep score (0-100) each night using Garmin Vivosmart 5 devices.

CONTACTS AND LOCATIONS:
Overall Officials: Collin Tukuitonga, Sir. Dr., Principal Investigator — University of Auckland, New Zealand
Locations (1):
- University of Auckland, Auckland, Niue

IPD SHARING:
Plan to Share IPD: Yes
Data that can be shared unconditionally underpinning the published research articles will be made available to other researchers at the time of publication, and data will be linked via the article DOI. Data that cannot be unconditionally shared upon publication owing to confidentiality or data protection requirements will be identified as such and a contact email will be provided in relevant publications for data access enquiries by other researchers.
  It is expected that demographic data of people at the study sites (family size and composition, basic socioeconomic indicators) may contain personally identifiable information and location data. All such data will be removed prior to storage on online data repositories and therefore will be available to be publicly shared at the time of publication of manuscripts.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the time of publication.
URL: http://reflect.org.nz

REFERENCES:
- See also: Related Info — http://reflect.org.nz